CLINICAL TRIAL: NCT01080365
Title: A Single Dose Bioequivalence Study Comparing The Commercial Tablet Formulation To The Clinical Tablet Of Bosutinib In Healthy Subjects
Brief Title: Study Comparing Two Different Tablet Formulations Of Bosutinib Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-1120; B1871016
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Commercial Tablet
  Interventions: Drug: SKI-606 (Bosutinib)
- 2 (Experimental): Clinical Tablet
  Interventions: Drug: SKI-606 (Bosutinib)

INTERVENTIONS:
Drug: SKI-606 (Bosutinib) — 500 mg commercial formulation film coated tablet, administered once daily
  Other Names: Bosutinib
  Arms: 1
Drug: SKI-606 (Bosutinib) — 500 mg (5 ×100 mg) phase 3 formulation film coated tablets, administered orally once daily
  Other Names: Bosutinib
  Arms: 2

SUMMARY:
Study comparing 2 formulations of bosutinib in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential age 18 to 50 years

Exclusion Criteria:

* Any clinically significant medical condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics, as measured by Cmax, AUC, tmax, t1/2 | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tacoma, Washington, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A4-1120&StudyName=Study%20Comparing%20Two%20Different%20Tablet%20Formulations%20Of%20Bosutinib%20Under%20Fed%20Conditions